CLINICAL TRIAL: NCT00135512
Title: An Open-Label, Multi-Center, Phase II Study Evaluating the Safety and Efficacy of 323U66 SR in Patients With Depression
Brief Title: Study Of 323U66 SR In Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK1102364
Record Dates: First submitted 2005-08-24; First posted 2005-08-26 (Estimated); Results first posted 2019-02-01 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2018-08

CONDITIONS: Depressive Disorder
Keywords: MDD
MeSH Terms: conditions — Depressive Disorder | interventions — Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: bupropion hydrochloride — Study drug

SUMMARY:
This study was designed to evaluate the efficacy and safety in major depressive disorder patients.

ELIGIBILITY:
Inclusion criteria:

* Met DSM-IV-TR criteria for major depressive disorder for their current episode for at least 8 weeks prior to screening visit.
* Must give a written informed consent. But if the patient is under 20, both the patient himself/herself and his/her proxy consenter must give written informed consent.
* Must have rating scores as outlined.

Exclusion criteria:

* Current or past history of seizure disorder or brain injury.
* Current or past history of anorexia or bulimia nervosa.
* History of manic episode.
* Past or current DSM- IV-TR diagnosis of schizophrenia or other psychotic disorder.
* Diagnosis of substance abuse (alcohol or drug) by the DSM-IV-TR criteria.
* Pregnant, possibly pregnant or lactating.
* Must not be suicidal.
* Blood pressure of SBP>160mmHg, DBP>100mmHg.
* History or complication of cancer or malignant tumour.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 234 (Actual)
Dates: Start 2004-12-01 (Actual); Primary Completion 2007-05-28 (Actual); Study Completion 2007-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- Japan (6):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Tokyo
- GSK Investigational Site

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 01 December 2004 to 28 May 2007, total of 234 participants with major depressive disorder were randomized at 36 centers in Japan.
Pre-assignment Details: During the screening (1 week), participants received Dose Level 1; bupropion sustained release (SR) 100 milligrams (mg) placebo tablet once daily in the morning.
Groups:
- Bupropion SR: During treatment period, participants received Dose Level 2; bupropion SR 100 mg tablets once daily for 1 week in the morning and then the Dose Level 3; bupropion SR 100 mg tablets twice daily (BID; morning and evening) for the next 1 week of the treatment phase. If no problems were observed in tolerability with insufficient efficacy, then Dose Level 4; bupropion SR 150 mg tablets BID for 6 weeks was administered. Dose reduction back to Dose Level 3 was allowed in participants judged by the investigator to have a safety concern after dose increase to Dose Level 4 and dose adjustment between Dose Levels 3 and 4 was to be chosen optionally. If no tolerability issues were observed at Week 8 of treatment phase, the treatment continued up to a maximum of 52 weeks. One tablet was administered per dose during each dose level.
Period: Overall Study
Arm/Group | Bupropion SR
Started | 234
Completed | 111
Not Completed | 123
Not completed — Adverse Event | 56
Not completed — Lack of Efficacy | 25
Not completed — Other | 42

BASELINE CHARACTERISTICS:
Population: Full analysis set was defined as all participants who entered treatment phase, except those who met any of the following criteria: did not satisfy the eligible disease criterion, received no dose of the investigational product and no observation data on post-treatment efficacy.
Groups:
- Bupropion SR: During treatment period, participants received Dose Level 2; bupropion SR 100 mg tablets once daily for 1 week in the morning and then the Dose Level 3; bupropion SR 100 mg tablets BID; morning and evening for the next 1 week of the treatment phase. If no problems were observed in tolerability with insufficient efficacy, then Dose Level 4; bupropion SR 150 mg tablets BID for 6 weeks. Dose reduction back to Dose Level 3 was allowed in participants judged by the investigator to have a safety concern after dose increase to Dose Level 4 and dose adjustment between Dose Levels 3 and 4 was to be chosen optionally. If no tolerability issues were observed at Week 8 of treatment phase, the treatment continued up to a maximum of 52 weeks. One tablet was administered per dose during each dose level.
Arm/Group | Bupropion SR
Number analyzed (Participants) | 232
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.1 (10.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101
  Male | 131
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race data for 231 participants is presented and race for 1 participant was unknown.
  Participants
    American Indian or Alaska Native | 0
    Asian | 231
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 0
    More than one race | 0
    Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Montgomery-Asberg Depression Rating Scale (MADRS) Total Score at Week 8 in Observed Cases
Description: The MADRS is a semi-structured interview rating scale for depression that assesses 10 symptoms. The scale is composed of 10 questions (1, apparent sadness; 2, reported sadness; 3, inner tension; 4, reduced sleep; 5, reduced appetite; 6, concentration difficulties; 7, lassitude; 8, inability to feel; 9, pessimistic thoughts; 10, suicidal thoughts) with a fixed 7 point scale (0, no depression; 60, severely depressed). Total score ranges from 0-60. A higher score indicates more depressive symptoms. MADRS Response was defined as a reduction in MADRS score from Baseline. Change from Baseline in the total score was calculated as the value at Week 8 minus the value at Baseline. Baseline was defined as value at Week 0.
Time Frame: Baseline (Week 0) and Week 8
Population: Full analysis set was used.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Bupropion SR
Number analyzed (Participants) | 232
Score on a scale | -16.8 (8.43)

2. Secondary Outcome: Change From Baseline in the MADRS Total Score at Week 52 in Observed Cases
Description: The MADRS is a semi-structured interview rating scale for depression that assesses 10 symptoms. The scale is composed of 10 questions (1, apparent sadness; 2, reported sadness; 3, inner tension; 4, reduced sleep; 5, reduced appetite; 6, concentration difficulties; 7, lassitude; 8, inability to feel; 9, pessimistic thoughts; 10, suicidal thoughts) with a fixed 7 point scale (0, no depression; 60, severely depressed). Total score ranges from 0-60. A higher score indicates more depressive symptoms. MADRS Response was defined as a reduction in MADRS score from Baseline. Change from Baseline in the total score was calculated as the value at Week 52 minus the value at Baseline. Baseline was defined as value at Week 0.
Time Frame: Baseline (Week 0) and Week 52
Population: Full analysis set was used.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Bupropion SR
Number analyzed (Participants) | 232
Score on a scale | -24.6 (8.34)

3. Secondary Outcome: Change From Baseline in the Hamilton Depression Rating Scale (HAM-D; 17 Items) Total Score at Weeks 8 and 52 in Observed Cases
Description: Each item was rated on either a 3-point scale (0 to 2; 8 questions) or a 5-point scale (0 to 4; 9 questions), with higher scores indicating greater symptom severity. The total score was calculated by summing the individual response scores. Total score ranged from 0 to 52. The following symptoms were rated on a 5-point scale (0-4): depressed mood, low self-esteem (guilt), suicidal thoughts, work and interests, psychomotor retardation, psychomotor agitation, anxiety (psychic), anxiety (somatic), and hypochondriasis (somatization). The following symptoms were rated on a 3-point scale (0-2): insomnia (initial), insomnia (middle), insomnia (late), gastrointestinal symptoms (appetite), somatic symptoms (general), sexual disturbances, insight, and weight loss. Change from Baseline in the total score was calculated as the score at Week 8 and 52 minus the score at Baseline. Baseline was defined as value at Week 0.
Time Frame: Baseline (Week 0) and Week 8, 52
Population: Full analysis set was used.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Bupropion SR
Number analyzed (Participants) | 232
Score on a scale
  Week 8 | -11.8 (6.06)
  Week 52 | -17.3 (6.38)

4. Secondary Outcome: Percentage of Participants Who Were Clinical Global Impression Global Improvement (CGI-I) Responders at Weeks 8 and 52 in Observed Cases
Description: The CGI-I scale was used to rate improvement in the participant's condition (benefits) since Baseline using the following 7-point scale: 1: very much improved, 2: much improved, 3: minimally improved, 4: not changed, 5: minimally worse, 6: much worse and 7: very much worse. A responder was defined as "very much improved" or "much improved".
Time Frame: Week 8, 52
Population: Full analysis set was used.
Measure: Number (95% Confidence Interval); unit: Percentage of participant
Arm/Group | Bupropion SR
Number analyzed (Participants) | 232
Percentage of participant
  Week 8 | 68.7 [61.0 to 75.6]
  Week 52 | 89.0 [81.6 to 94.2]

5. Secondary Outcome: Change From Baseline in CGI Severity of Illness (CGI-SI) at Weeks 8 and 52 in Observed Cases
Description: CGI-SI was assessed on an 8-grade scale: 0, not assessed; 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill and 7, among the most extremely ill. Higher score indicated severely ill. CGI-SI was assessed by the investigator. The change from Baseline in CGI-SI score was calculated as the score at Weeks 8 and 52 minus the score at Baseline. Baseline was defined as value at Week 0.
Time Frame: Baseline (Week 0) and Week 8, 52
Population: Full analysis set was used.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Bupropion SR
Number analyzed (Participants) | 232
Score on a scale
  Week 8 | -1.3 (0.98)
  Week 52 | -2.3 (1.16)

6. Secondary Outcome: Change From Baseline in the Sheehan Disability Scale (SDISS) Total Score at Weeks 8 and 52 in Observed Cases
Description: SDISS is a composite of 3 self-rated items designed to measure the extent to which 3 major sectors in the participant's life are impaired by panic, anxiety, phobic, or depressive symptoms. The participant rates the extent to which his or her (1) work, (2) social life or leisure activities, and (3) home life or family responsibilities were impaired by his or her symptoms on a 10-point visual analog scale. To get a total score, 3 individual scores were added and the total score ranged from "0 = unimpaired" to "30 = highly impaired". Higher scores indicate worsening. The change from Baseline in SDISS total score was calculated as the score at Weeks 8 and 52 minus the score at Baseline. Baseline was defined as value at Week 0.
Time Frame: Baseline (Week 0) and Week 8, 52
Population: Full analysis set was used.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Bupropion SR
Number analyzed (Participants) | 232
Score on a scale
  Week 8 | -5.0 (5.54)
  Week 52 | -9.7 (7.31)

7. Secondary Outcome: Change From Baseline in the Motivation Energy Inventory Short Form (MEI-SF) Total Score at Weeks 8 and 52 in Observed Cases
Description: The MEI-SF (18 questions) was used to measure the reductions in mental energy, physical energy and social motivation. Minimal clinically important differences were estimated as 0.5 standard deviations or 7.5 points. All items use either a 7-level (0 to 6) or 5-level (0 to 4) response scale; items with a 5-level response scale were rescaled to 7-levels and items were reverse-scored as necessary such that higher scores represent higher health-related quality of life (HRQoL) total score ranges from 0 to 108 points. Recall period was past week prior to administration. The change from Baseline in MEI-SF total score was calculated as the score at Weeks 8 and 52 minus the score at Baseline. Baseline was defined as value at Week 0.
Time Frame: Baseline (Week 0) and Week 8, 52
Population: Full analysis set was used.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Bupropion SR
Number analyzed (Participants) | 232
Score on a scale
  Week 8 | 15.2 (15.51)
  Week 52 | 26.7 (20.54)

ADVERSE EVENTS:
Time Frame: All adverse events (AE) and serious adverse events (SAE) were reported up to Week 52.
Description: All participants who had participated in the study and had received at least 1 dose of the investigational product were included in the safety population and were used for reporting non-SAE and SAE.
Arm/Group | Bupropion SR
All-Cause Mortality (participants affected / at risk) | 1/233
Serious Adverse Events (participants affected / at risk) | 14/233
Other Adverse Events (participants affected / at risk) | 210/233
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bupropion SR (N=233)
Depression (Psychiatric disorders) | 3
Suicidal ideation (Psychiatric disorders) | 1
Back injury (Injury, poisoning and procedural complications) | 1
Intentional misuse (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Grand mal convulsion (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Gastroenteritis bacterial (Infections and infestations) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1
Genital haemorrhage (Reproductive system and breast disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Death (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bupropion SR (N=233)
Nasopharyngitis (Infections and infestations) | 85
Thirst (General disorders) | 42
Nausea (Gastrointestinal disorders) | 26
Headache (Nervous system disorders) | 22
Depression (Psychiatric disorders) | 17
Dizziness (Nervous system disorders) | 16
Abdominal pain upper (Gastrointestinal disorders) | 14
Constipation (Gastrointestinal disorders) | 14
Diarrhoea (Gastrointestinal disorders) | 14
Stomach discomfort (Gastrointestinal disorders) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.